CLINICAL TRIAL: NCT05752864
Title: The Effects of Sacroiliac Joint Manual Therapy on Autonomic Nervous System and Lower Abdominal Pain in Women in Their 20s With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyun-Joong Kim, Doctor, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYU 2023-01-002-002
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spine manual therapy of sacroiliac joint (Experimental): The group which treats spine manual therapy of sacroiliac joint
  Interventions: Behavioral: spine manual therapy
- Superficial heat therapy (Active Comparator): Group treated with superficial heat therapy for 20 minutes
  Interventions: Device: Superficial heat therapy

INTERVENTIONS:
Behavioral: spine manual therapy — The manual treatment method applied to the sacroiliac joint used high-velocity, low amplitude (HVLA).
  Arms: spine manual therapy of sacroiliac joint
Device: Superficial heat therapy — In the physical therapy used in this study, it was applied for 20 minutes using conventionally used superficial heat therapy.
  Arms: Superficial heat therapy

SUMMARY:
Disorders of the autonomic nervous system are considered another possible cause of dysmenorrhea. spinal manual threapty is acting on the parasympathetic and sympathetic nerves.

The sacrum affects all vertebrae, which affects the position of this bone, is thought to have a lot to do with dysmenorrhea.

In this study, by applying spinal manual threapty threapty to the sacroiliac joint in women in their 20s with primary dysmenorrhea, we tried to present an effective treatment method by evaluating the function of the autonomic nervous system and confirming the occurrence of pain in the lower abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 20-29
* Regular menstrual cycle (24-32 days)
* Those who have had symptoms of primary dysmenorrhea for at least 1 year
* Those who have lower back pain symptoms related to menstrual pain of 5 or higher on the Visual Analysis Scale (VAS)
* The body mass index is between 20-30
* Positive reaction to Gillet test

Exclusion Criteria:

* pelvic inflammatory disease
* uterine fibroids, polycystic ovary syndrome. Those with gynecological findings such as endometriosis
* Those who have used an intrauterine contraceptive device
* Those who took birth control pills or nonsteroidal anti-inflammatory drugs at the time of the experiment

Ages: 20 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | Change from baseline after intervention at 4 weeks, follow-up at 4 weeks
  Autonomic nervous system balance tester (SA3000new, Medicore Co. Korea) was used. The subjects placed electrodes on three areas (left arm, left leg, right leg) while lying down and performed for 3 minutes.

SECONDARY OUTCOMES:
Visual analog scale | Change from baseline after intervention at 4 weeks, follow-up at 4 weeks
  On a line consisting of 10 cm, 0 at either end represents 'no pain' and 10 represents 'worst pain'.
Pressure pain threshold | Change from baseline after intervention at 4 weeks, follow-up at 4 weeks
  The test determines the amount of pressure over a given area in which a steadily increasing nonpainful pressure stimulus turns into a painful pressure sensation. With the participant seated comfortably, the examiner identified the sacroiliac joint and applied pressure with the algometer perpendicular to the skin surface until the participant made an "Ah" sound.
  * Lower pressure pain thresholds indicate higher sensitivity to pressure and a lower pain tolerance.
  * Higher pressure pain thresholds suggest lower sensitivity and a higher pain tolerance.
Menstrual distress questionnaire | Change from baseline after intervention at 4 weeks, follow-up at 4 weeks
  The Menstrual Distress Questionnaire (MDQ) is a standard method for measuring cyclical menstrual cycle symptoms. The MDQ can differentiate between cyclical and non-cyclical changes in somatic symptoms, mood and behavior, and arousal.
  -The measured scores range from 0 to 185; higher scores indicate severe dysmenorrhea symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sungeon Park, Ph.D candidate, Principal Investigator — The wells neuropain clinic
Locations (1):
- The wells neuropain clinic, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes